CLINICAL TRIAL: NCT02765152
Title: Effects of Training Rhythmic and Discrete Aiming Movements on the Upper Limb Control and Functionality After Stroke: Randomized Controlled Trial
Brief Title: Effects of Training Rhythmic and Discrete Aiming Movements on Arm Control and Functionality After Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Cidade de Sao Paulo (Other)
Responsible Party: Principal Investigator, Renata Morales Banjai, Principal Investigator, Universidade Cidade de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Universidade Cidade Sao Paulo
Record Dates: First submitted 2016-04-19; First posted 2016-05-06 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Stroke
Keywords: exercise; rhythmic movement; discrete movement
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Conventional Physical Therapy (Active Comparator): Usual therapy: joint mobility exercises, stimulating joint movement of the main active components of the upper limb; major muscle groups stretching, especially in the affected muscles by tone impairment; manual resistance training according to the degree of the patient's muscle strength, prioritizing the functional specificity of the upper limb, so the majority of the exercises will be held in open chain; motor coordination exercises, unilateral and bilateral motor tasks as well as task-oriented training of the upper limb with a focus on functional tasks.
  Interventions: Other: Conventional Physical Therapy
- discrete movement training group (Experimental): Aiming movements training with the affected upper limb (unilateral training) or both limbs (bilateral training) on the surface of a table. The starting point of the movement and its target are predetermined. Targets will be placed in different directions and distances from the starting point and the therapist ask for variations on speed and assistance, if necessary.
  Interventions: Other: Discrete movement training group
- rhythmic movement training group (Experimental): Aiming movements training with the affected upper limb (unilateral training) or both limbs (bilateral training) on the surface of a table. The movement begins in a predetermined starting point, directed to a target and returns to the starting point. This activity is performed several times with rhythmic movements. Targets will be placed in different directions and distances from the starting point and the therapist ask for variations on speed and assistance, if necessary.
  Interventions: Other: Rhythmic movement training group

INTERVENTIONS:
Other: Conventional Physical Therapy — Combination of joint mobility exercises, specific exercises for muscle strength and motor coordination exercises, unilateral and bilateral motor tasks as well as task-oriented training of the upper limb with a focus on functional tasks. Patients will receive 10 sessions of treatment over a period of five weeks (two sessions/week)
  Arms: Conventional Physical Therapy
Other: Discrete movement training group — Aiming movements training with the affected upper limb (unilateral training) or both limbs (bilateral training) on the surface of a table. The starting point of the movement and its target are predetermined. Targets will be placed in different directions and distances from the starting point and the therapist ask for variations on speed and assistance, if necessary.
  Arms: discrete movement training group
Other: Rhythmic movement training group — Aiming movements training with the affected upper limb (unilateral training) or both limbs (bilateral training) on the surface of a table. The movement begins in a predetermined starting point, directed to a target and returns to the starting point. This activity is performed several times with rhythmic movements. Targets will be placed in different directions and distances from the starting point and the therapist ask for variations on speed and assistance, if necessary.
  Arms: rhythmic movement training group

SUMMARY:
The purpose of this study is to verify the additional effects of rhythmic specific training, discrete specific training additional to conventional therapy on the upper limb after chronic stroke subjects on the outcomes: motor control and functionality.

DETAILED DESCRIPTION:
Seventy-five patients will be randomized into three groups to receive conventional therapy, consisting of a combination of mobility exercises joint, muscle stretching, strength training, motor coordination exercises, unilateral and bilateral motor tasks as well as oriented tasks training upper limb with a focus on functional tasks. The other groups will receive additional intervention consisting of aiming movement practice according two different protocols: discrete movements to targets placed in different directions and distances; and rhythmic movements also to targets placed in different directions and distances. Both additional interventional interventions will be conducted for 30 minutes over a 5 week-period (total: 10 sessions).

Clinical outcomes (motor control), functional and kinematic will be collected at baseline and at five weeks. Functional results will be collected at the beginning, after 5 weeks and 3 months after randomization. Data will be collected by a blinded assessor on patients' allocation group. All statistical analyzes will be carried out following the principles of intention to treat analysis and differences between groups will be performed using linear mixed models.

ELIGIBILITY:
Inclusion criteria:patients who participate in the survey, adult stroke survivors (>18 years), with primary diagnosis of first-ever unilateral stroke (ischaemic or haemorrhagic), stroke experienced > 6 months prior to study enrollment and score ≥ 20 on the Folstein Mini Mental Status Examination.

Exclusion criteria: patients with excessive pain in the paretic hand, arm or shoulder excessive spasticity at the paretic elbow and wrist as defined as a score of 4 on the Modified Ashworth Spasticity Scale and upper limb comorbidities that could limit their functional recovery (e.g., arthritis, pain, other neurological disorders).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-06 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Stroke Impact Scale (SIS) | Five weeks after randomization and 3 months after randomization
  Functionality: questionnaire which evaluates functionality. In this study will be evaluated four areas (arm muscle strength, hand function, activities of daily living and social participation)(Duncan et al., 1999). Each domain is scored from 1 to 5 (1 point corresponds to the worst possible outcome and 5 points to the best result). For the four areas the lowest possible score is 28 points and the highest is 125 points.

SECONDARY OUTCOMES:
Motor Activity Log (MAL) | Five weeks and 3 months after randomization
  Arm function: individuals are asked to rate Quality of Movement (QOM) and Amount of Movement (AOM) during 30 daily functional tasks (original MAL) (Uswatte et al., 2005).
  Items scored on a 6-point ordinal scale, where 0 corresponds to the weaker arm was not sued at all for that activity (never). Patients with a score 5 show the ability to use the weaker arm for that activity was as good as before the stroke (normal).
Fugl-Meyer Assessment Scale | Five weeks after randomization
  Motor control: this scale assesses sensorimotor function of upper limb, with score 0-66 points with scores 0-66 points for motor function and 0-126 points for sensory-motor function (Fugl-Meyer, 1975). A higher score is better motor function.

OTHER OUTCOMES:
kinematics assessment | Five weeks after randomization
  Functional capacity: It will be used an experimental apparatus that analyzes the motor behavior the aiming movement (Ribeiro et al., 2014). They will evaluate the movement time (measured in milliseconds), reaction time (in milliseconds) and smoothness (expressed in units of motion). The movement time is the time interval between the beginning and the end of the movement. Reaction time is defined as the time between the start of the imperative stimulus to the beginning of the movement. The smoothness is evaluated by computing the number of times the acceleration zero crossing (positive to negative and vice versa). The resultant variable error (in centimeters) is a measure of variability for both the medial-lateral direction as anteroposterior, assessing the accuracy to hit the target.
Grip strength | Five weeks after randomization
  Body function and structure: it will measure the strength of grip and pinch through dynamometer. The results will be presented in kilogram-force (Kgf) (Mathiowetz et al., 1985)
Modified Ashworth Spasticity Scale | Five weeks after randomization
  Body function and structure: they will be assessed flexors elbow, wrist and fingers, and forearm pronators. A measurement scale from 0 to 4 points, with 0 representing normal muscle tone and 4 is the highest possible degree of spasticity (Bohannon and Smith, 1987)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra R Alouche, PhD, Study Director — Universidade Cidade São Paulo
Locations (1):
- Universidade Cidade de Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cauraugh JH, Summers JJ. Neural plasticity and bilateral movements: A rehabilitation approach for chronic stroke. Prog Neurobiol. 2005 Apr;75(5):309-20. doi: 10.1016/j.pneurobio.2005.04.001. PMID 15885874
- [Background] Naghdi S, Ansari NN, Mansouri K, Hasson S. A neurophysiological and clinical study of Brunnstrom recovery stages in the upper limb following stroke. Brain Inj. 2010;24(11):1372-8. doi: 10.3109/02699052.2010.506860. PMID 20715900
- [Background] Harris JE, Eng JJ. Paretic upper-limb strength best explains arm activity in people with stroke. Phys Ther. 2007 Jan;87(1):88-97. doi: 10.2522/ptj.20060065. Epub 2006 Dec 19. PMID 17179441
- [Background] Faria-Fortini I, Michaelsen SM, Cassiano JG, Teixeira-Salmela LF. Upper extremity function in stroke subjects: relationships between the international classification of functioning, disability, and health domains. J Hand Ther. 2011 Jul-Sep;24(3):257-64; quiz 265. doi: 10.1016/j.jht.2011.01.002. Epub 2011 Mar 21. PMID 21420279
- [Background] Sirtori V, Corbetta D, Moja L, Gatti R. Constraint-induced movement therapy for upper extremities in stroke patients. Cochrane Database Syst Rev. 2009 Oct 7;(4):CD004433. doi: 10.1002/14651858.CD004433.pub2. PMID 19821326
- [Background] Liepert J. Evidence-based therapies for upper extremity dysfunction. Curr Opin Neurol. 2010 Dec;23(6):678-82. doi: 10.1097/WCO.0b013e32833ff4c4. PMID 20852418
- [Background] Ada L, O'Dwyer N, O'Neill E. Relation between spasticity, weakness and contracture of the elbow flexors and upper limb activity after stroke: an observational study. Disabil Rehabil. 2006 Jul 15-30;28(13-14):891-7. doi: 10.1080/09638280500535165. PMID 16777777
- [Background] Oujamaa L, Relave I, Froger J, Mottet D, Pelissier JY. Rehabilitation of arm function after stroke. Literature review. Ann Phys Rehabil Med. 2009 Apr;52(3):269-93. doi: 10.1016/j.rehab.2008.10.003. Epub 2009 Apr 9. English, French. PMID 19398398
- [Background] Cauraugh JH, Lodha N, Naik SK, Summers JJ. Bilateral movement training and stroke motor recovery progress: a structured review and meta-analysis. Hum Mov Sci. 2010 Oct;29(5):853-70. doi: 10.1016/j.humov.2009.09.004. Epub 2009 Nov 18. PMID 19926154
- [Background] van Delden AE, Peper CE, Beek PJ, Kwakkel G. Unilateral versus bilateral upper limb exercise therapy after stroke: a systematic review. J Rehabil Med. 2012 Feb;44(2):106-17. doi: 10.2340/16501977-0928. PMID 22266762
- [Background] Chang JJ, Tung WL, Wu WL, Huang MH, Su FC. Effects of robot-aided bilateral force-induced isokinetic arm training combined with conventional rehabilitation on arm motor function in patients with chronic stroke. Arch Phys Med Rehabil. 2007 Oct;88(10):1332-8. doi: 10.1016/j.apmr.2007.07.016. PMID 17908578
- [Background] Smits-Engelsman BC, Swinnen SP, Duysens J. The advantage of cyclic over discrete movements remains evident following changes in load and amplitude. Neurosci Lett. 2006 Mar 20;396(1):28-32. doi: 10.1016/j.neulet.2005.11.001. Epub 2005 Dec 2. PMID 16326008
- [Background] Duncan PW, Wallace D, Lai SM, Johnson D, Embretson S, Laster LJ. The stroke impact scale version 2.0. Evaluation of reliability, validity, and sensitivity to change. Stroke. 1999 Oct;30(10):2131-40. doi: 10.1161/01.str.30.10.2131. PMID 10512918
- [Background] Uswatte G, Taub E, Morris D, Vignolo M, McCulloch K. Reliability and validity of the upper-extremity Motor Activity Log-14 for measuring real-world arm use. Stroke. 2005 Nov;36(11):2493-6. doi: 10.1161/01.STR.0000185928.90848.2e. Epub 2005 Oct 13. PMID 16224078
- [Background] Fugl-Meyer AR, Jaasko L, Leyman I, Olsson S, Steglind S. The post-stroke hemiplegic patient. 1. a method for evaluation of physical performance. Scand J Rehabil Med. 1975;7(1):13-31. PMID 1135616
- [Background] Ribeiro Coqueiro P, de Freitas SM, Assuncao e Silva CM, Alouche SR. Effects of direction and index of difficulty on aiming movements after stroke. Behav Neurol. 2014;2014:909182. doi: 10.1155/2014/909182. Epub 2014 Jan 28. PMID 24803738
- [Background] Mathiowetz V, Kashman N, Volland G, Weber K, Dowe M, Rogers S. Grip and pinch strength: normative data for adults. Arch Phys Med Rehabil. 1985 Feb;66(2):69-74. PMID 3970660
- [Background] Bohannon RW, Smith MB. Interrater reliability of a modified Ashworth scale of muscle spasticity. Phys Ther. 1987 Feb;67(2):206-7. doi: 10.1093/ptj/67.2.206. PMID 3809245